CLINICAL TRIAL: NCT03088982
Title: Running Title: The Patient's Pain Seems to be a Reliable Risk Factor for Decompensation Among Multimorbid Patients in Residential Care.
Brief Title: Preventing Decompensation Among Multimorbid Outpatients in Residential Care. A Cohort Study With a Six-month Follow-up.
Acronym: FDPM
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Collaborators: ERCR SPURBO (Other); Unité INSERM 1078, SFR 148 ScInBioS, Brest (Unknown)
Responsible Party: Sponsor
Other Study IDs: FDPM - 05122011
Record Dates: First submitted 2017-03-14; First posted 2017-03-24 (Actual); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Multimorbidity
Keywords: Family Medicine; multimorbidity; prevention
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lanmeur multimorbid patients: All multimorbid patients who met 12 FPs in the Lanmeur residential care home in the county of Finistere (in north-west France) from July 2014 to December 2014. These FPs were drawn from those physicians associated with the Lanmeur residential care home.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — FPs who had agreed to participate worked according to the following plan: first, the multimorbid patient was asked to give his/her consent to participate in the study once the terms had been explained to him/her. After that, FPs completed a questionnaire about their patient.
  The purpose of this questionnaire was to explore potential decompensation risk factors within the themes and subthemes of multimorbidity.

SUMMARY:
Background :The European General Practitioners Research Network (EGPRN) designed and validated a comprehensive definition of multimorbidity using a systematic literature review and qualitative research throughout Europe. This survey assessed which criteria in the EGPRN concept of multimorbidity could detect decompensating patients in residential care within a primary care cohort at a 6-month follow-up.

Method: Family Physicians included all multimorbid patients encountered in their residential care homes from July to December 2014. Inclusion criteria were those of the EGPRN definition of Multimorbidity. Exclusion criteria were patients under legal protection and those unable to complete the 2-year follow-up. Decompensation was defined as the occurrence of death or hospitalization for more than seven days. Statistical analysis was undertaken with uni- and multivariate analysis at a 6-month follow-up using a combination of approaches including both automatic classification and expert decision making. A Multiple Correspondence Analysis (MCA) and a Hierarchical Clustering on Principal Components (HCPC) confirmed the consistency of the results. Finally a logistic regression was performed in order to identify and quantify risk factors for decompensation.

DETAILED DESCRIPTION:
The concept of multimorbidity was first published in 1976. Multimorbidity has been defined by the World Health Organization (WHO) as people being affected by two or more chronic health conditions. Multimorbidity is a very interesting and challenging concept particularly for Family Medicine (FM), given the increasing prevalence of chronic illness in an aging population across all developed countries. It is closely related to a global or comprehensive view of the patient, which is a core competency of FM, as defined, for instance, by the World Organization of National Colleges, Academies and Academic Associations of General Practitioners/Family Physicians (WONCA). It is a global 'functional' view (useful for Long-Term Care) versus a 'disease' centered point of view (useful for acute care).

The European General Practice Research Network (EGPRN) has created a research agenda specifically designed for methodological and instrumental research, which includes the development of primary care epidemiology, focusing on patient-centered health. A comprehensive definition of the concept of multimorbidity (i.e. one which is both understandable and usable for further collaborative research) was an important objective for this research network. The objective was to help researchers in FM to investigate the complexity of patients' conditions and their overall impact on patients' health. This concept of multimorbidity could be an additional tool for Family Physicians (FPs), enabling them to prevent decompensation.

A research team, including 9 national groups, all active within the EGPRN, has created a research community for the purpose of clarifying the concept of multimorbidity for FM throughout Europe. This group produced a comprehensive definition of the concept of multimorbidity through a systematic review of literature. This concept was translated into most European languages for use in further collaborative research. Finally, it was validated using qualitative research throughout Europe and a specific research agenda was issued. The EGPRN concept of multimorbidity included a set of different variables assessing patients' multimorbidity, multimorbidity modulating factors and multimorbidity consequences.

Decompensation (i.e. death or hospitalization in acute care) is a challenge for FM as FPs, being familiar with their patient's health status, could miss tiny factors which, if noticed, could help to prevent decompensation. A predictive model that could be integrated into their clinical practice could help them to prevent decompensation and avoid serious health outcomes for their patients. The EGPRN concept of multimorbidity was considered highly suitable for a purpose such as this. It could lead to a usable model for preventing decompensation.

The French population is aging, with one in three people over 60 years of age in 2050. Consequently, the number of dependent patients, some requiring institutionalization in Care homes (CHs), is growing. Patients residing in CHs are included in the EGPRN definition of multimorbidity. In France, as in most European countries, patients in residential care are treated by FPs.

The purpose of this research was to assess which criteria in the EGPRN concept of multimorbidity could detect decompensating patients in residential care within a primary care cohort at a 6-month follow-up.

ELIGIBILITY:
Inclusion criteria were patients meeting the criteria for the definition of multimorbidity according to the EGPRN definition: any combination of chronic disease with at least another disease (acute or chronic) or a bio psychosocial factor (associated or not) or somatic risk factor.

Exclusion criteria were patients not meeting the criteria of the definition of multimorbidity, the inability to follow the study over time, patients on legal protection, patients for whom survival was estimated at less than three months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population included all multimorbid patients (according to the EGPRN definition of multimorbidity) who met 12 FPs in the Lanmeur residential care home in the county of Finistere (in north-west France) from July 2014 to December 2014. These FPs were drawn from those physicians associated with the Lanmeur residential care home.
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Evaluation of the multimorbidity criteria | 6 months
  The purpose of this research was to assess which criteria in the EGPRN concept of multimorbidity could detect decompensating patients in residential care within a primary care cohort at a 6-month follow-up.

IPD SHARING:
Plan to Share IPD: No